CLINICAL TRIAL: NCT01041820
Title: Critical Periods of Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Krista Casazza, Krista R. Casazza PhD, RD/Assistant Professor, UAB, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F090904001
Record Dates: First submitted 2009-12-30; First posted 2010-01-01 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Metabolism
Keywords: exercise; bone marrow adipose tissue; bone mineral density; Children in the intervention condition will complete a supervised physical activity program 3 days/wk for 10 weeks; Control treatment will be provided no intervention; All participants will be instructed not to change their current dietary habits during the study period.
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise group (Experimental): Children will participate in a 10-week moderate to vigorous exercise program
  Interventions: Behavioral: Exercise
- non-exercising (No Intervention): Participants will receive no intervention

INTERVENTIONS:
Behavioral: Exercise — Children will be exposed to a 10-week exercise intervention
  Arms: Exercise group

SUMMARY:
Early childhood (~3-7 years of age) is an important window for determining body composition trajectory and may be a critical period for the development of tissue partitioning patterns that influence obesity risk. As adiposity accelerates during this critical period, deposition/ preservation of fat stores may be sustained at the 'expense' of other tissues; i.e. energy homeostasis may be inherently biased toward fat gain. The type and amount of tissue mass accrued in early childhood has implications for metabolic profile, glucose/insulin homeostasis, hormone profile and resting energy expenditure.

The interplay between fat and bone deposition represents a physiologic trait enabling the body to choose between shuttling 'energy' towards accrual of a particular tissue. Plausibly the phenotype underlying obesity and diabetes risk may be determined by the differentiation of cell type (adipocyte, osteocyte, etc.) during this early stage of growth and development. In vitro studies demonstrate transdifferentiation under the influence of specific external stimuli, which can switch phenotypes toward other cell lineages. Further, rodent models have demonstrated that exposure to stimuli (exercise) early in life may prevent excess fat mass accrual in adulthood, even when the stimulus is later removed (animals are no longer exercising). Children's early experiences (engagement in physical activity vs. sedentary behavior) may 'environmentally induce' alterations in body composition and predispose individuals to obesity throughout life.

Aim 1. To examine the associations between body composition via DXA and objectively-measured physical activity/inactivity.

1. Hypothesis 1.1: There is a positive association between physical activity and bone mass.
2. Hypothesis 1.2: There is a positive association between sedentary behavior and total fat mass.

   Aim2. To examine the associations between adipose tissue distribution via MRI and objectively-measured physical activity/inactivity.
3. Hypothesis 2.1: There is an inverse association between physical activity and bone marrow adipose tissue.
4. Hypothesis 2.2: There is a positive association between sedentary behavior and bone marrow adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* children aged 3 to 7 years
* healthy, not under the care of a doctor
* not taking medications known to alter body composition or metabolism

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Association between exercise and bone marrow adipose tissue in children 3-7 years | 10 weeks of exercise

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Family Care Center, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama